CLINICAL TRIAL: NCT03874234
Title: A Randomized, Double-blind (Sponsor Unblinded), Placebo-controlled, First Time in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single (in Both Fed and Fasted States) and Repeat Doses of GSK3186899 in Healthy Participants
Brief Title: Safety, Tolerability and Pharmacokinetics (PKs) Investigation of GSK3186899 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated early following strategic review after emergence of nonclinical data with a non-GlaxoSmithKline asset.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 208436
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-05

CONDITIONS: Leishmaniasis
Keywords: Dose escalation phase; First time in human; Single ascending dose; Multiple ascending dose; GSK3186899
MeSH Terms: conditions — Leishmaniasis | interventions — GSK3186899

STUDY DESIGN:
Intervention Model Description: Subjects will receive escalating doses of GSK3186899 and placebo in Part A of the study. Subjects will receive repeat doses either of GSK3186899 or placebo in Part B of the study.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Subjects and Investigator will be blinded to the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: Subjects receiving GSK3186899 + placebo in Cohort 1 (Experimental): Subjects will receive 3 single ascending oral doses (SAD) of GSK3186899 and 1 dose of placebo as spray dried powder, under fasted conditions on Day 1 of cohort 1 in each of the four treatment periods. In each treatment period GSK3186899 and placebo will be administered in a 3:1 ratio. A wash out period of at least 10 days will be maintained between each treatment period.
  Interventions: Drug: GSK3186899; Drug: Placebo
- Part A: Subjects receiving GSK3186899 + placebo in Cohort 2 (Experimental): Subjects will receive 3 SAD of GSK3186899 and 1 dose of placebo as spray dried powder, under fasted conditions on Day 1 of cohort 2 in each of the four treatment periods. In each treatment period GSK3186899 and placebo will be administered in a 3:1 ratio. A wash out period of at least 10 days will be maintained between each treatment period.
  Interventions: Drug: GSK3186899; Drug: Placebo
- Part A: Subjects receiving GSK3186899 in Cohort 3 (Experimental): Subjects will receive GSK3186899 orally, under fasted condition and fed conditions on Day 1 of cohort 3 in each of the two treatment periods. There will be a wash out period of at least 10 days between each treatment period. A dose level will be determined based on the effect of food on the safety, tolerability and PK of a single dose of GSK3186899, with dose level selected from Cohorts 1 and 2.
  Interventions: Drug: GSK3186899
- Part B: Subjects receiving GSK3186899 (Experimental): Subjects will receive GSK3186899, orally, twice daily (BID) on Days 1 to 10. Subjects will receive each dose after either fed or fasted conditions. Part B will be initiated based on the review of all safety, tolerability and PK data from Part A.
  Interventions: Drug: GSK3186899
- Part B: Subjects receiving placebo (Placebo Comparator): Subjects will receive placebo, orally, BID on Days 1 to 10. Subjects will receive each dose after either fed or fasted conditions. Part B will be initiated based on the review of all safety, tolerability and PK data from Part A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3186899 — GSK3186899 will be available as white to slightly colored, spray dried powder in a bottle to be administered orally along with mixture of propylene glycol and water.
  Arms: Part A: Subjects receiving GSK3186899 + placebo in Cohort 1; Part A: Subjects receiving GSK3186899 + placebo in Cohort 2; Part A: Subjects receiving GSK3186899 in Cohort 3; Part B: Subjects receiving GSK3186899
Drug: Placebo — Placebo will be available as white to slightly colored, blend powder in a bottle to be administered orally along with mixture of propylene glycol and water.
  Arms: Part A: Subjects receiving GSK3186899 + placebo in Cohort 1; Part A: Subjects receiving GSK3186899 + placebo in Cohort 2; Part B: Subjects receiving placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and PK profile of single and repeat ascending doses of GSK3186899 in healthy subjects. This is a Phase 1 first time in human study, to investigate the effect of food on PK of GSK3186899. This study will consists of two parts. Part A (dose escalation phase) will be a single ascending, sequential cross-over design in cohorts 1, 2 and 3 of subjects. Cohort 1 and 2 will be 4-way cross-over which includes 4 dosing regimens of GSK3186899 and placebo (3:1 ratio) under fasted conditions. Cohort 3 will be 2-way cross-over which includes 2 treatment periods, 2 dosing regimens in fasted and fed conditions. In Part B (repeat dose escalation phase) subjects will be randomized to receive repeat doses of either GSK3186899 or placebo (3:1 ratio) in either fed or fasted conditions. Part B will be conducted based on the review of all safety, tolerability and PK data from Part A. The study duration includes screening, treatment periods and follow-up.

ELIGIBILITY:
Inclusion Criteria

* Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included only if the Investigator in consultation with the Medical Monitor (if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18.5 to 28 kilogram per square meter (kg/m^2) (inclusive).
* Male and/or female subjects: A male subject with a female partner of reproductive potential must agree to use contraception during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period. A female subject is eligible to participate if she is not a woman of childbearing potential (WONCBP).
* Capable of giving signed informed consent.

Exclusion Criteria

* History or presence of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Previous history of leishmaniasis.
* ALT >1.5* upper limit of normal (ULN).
* Bilirubin >1.5*ULN (isolated bilirubin >1.5*ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or past history of clinically significant gastritis or gastroduodenal ulcers or regular use of non-steroidal anti-inflammatory drugs (NSAID).
* ECG QT interval corrected for heart rate (QTc) >450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication, including herbal medications, NSAIDs, proton-pump inhibitors (PPIs) or anti-H2 antagonists within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longest) prior to dosing. Other concomitant medication may be considered on a case by case basis by the Investigator in consultation with the medical monitor.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within a 56-day period.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates participation in the study.
* Regular use of known drugs of abuse.
* Subjects with renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) with an age appropriate glomerular filtration rate (GFR) <=80 (mL/minute/1.73m^2).
* Presence of Hepatitis B surface antigen (HBsAg) or Positive Hepatitis C antibody test result at screening.
* Positive human immunodeficiency virus (HIV) antibody test.
* Positive pre-study drug/alcohol screen.
* Presence of clinically significant hematuria and/or proteinuria.
* Carbon monoxide levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 3 months prior to screening.
* Part A (Food effect) Cohort 3 only: Subject must have no dietary restrictions (example, lactose intolerance) or inability to eat an adapted standard meal (includes 35-40 percent fat content).
* Part A (Food effect) Cohort 3 only: History of gall bladder surgery or gall bladder removal, or history of an acute disease state (example, cholelithiasis) within 14 days prior to receiving the study treatment.
* Part B only: Early morning cortisol <420 nanomoles per liter (nmol/L) and inadequate response (rise of <250 millimoles per liter (mmol/L) from Baseline) to adrenocorticotropic hormone (ACTH) stimulation test at Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was 2-part study. Part A comprised of 3 Cohorts (Cohorts 1, 2 and 3); Part B comprised 3 cohorts (Cohorts 4, 5 and 6). Study was terminated after completion of Cohort 2, Period 3 of Part A following strategic review after emergence of nonclinical data with non-GlaxoSmithKline asset. Hence, no participants were enrolled in Cohort 2 Period 4 and Cohort 3 of Part A and in all Cohorts of Part B.
Pre-assignment Details: A total 25 participants were enrolled (Enrolled Population consisted of all participants who passed screening and entered the study) in this study (Part A: Cohort 1- 11 participants, Cohort 2- 14 participants). Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Groups:
- Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo: Participants in Part A Cohort 1 received a single dose of GSK3186899 30 milligram (mg) on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 60 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 120 mg on Day 1 in treatment Period 3; further followed by a single dose of Placebo on Day 1 in treatment Period 4. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg: Participants in Part A Cohort 1 received a single dose of GSK3186899 30 mg on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 60 mg on Day 1 in treatment Period 2; followed by a single dose of Placebo on Day 1 in treatment Period 3; further followed by a single dose of GSK3186899 300 mg on Day 1 in treatment Period 4. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg: Participants in Part A Cohort 1 received a single dose of GSK3186899 30 mg on Day 1 in treatment Period 1; followed by a single dose of Placebo on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 120 mg on Day 1 in treatment Period 3; further followed by a single dose of GSK3186899 300 mg on Day 1 in treatment Period 4. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg: Participants in Part A Cohort 1 received a single dose of Placebo on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 60 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 120 mg on Day 1 in treatment Period 3; further followed by a single dose of GSK3186899 300 mg on Day 1 in treatment Period 4. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo: Participants in Part A Cohort 2 received a single dose of GSK3186899 300 mg on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 600 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 800 mg on Day 1 in treatment Period 3; further followed by a single dose of Placebo on Day 1 in treatment Period 4. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7: Participants in Part A Cohort 2 received a single dose of GSK3186899 300 mg on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 600 mg on Day 1 in treatment Period 2; followed by a single dose of Placebo on Day 1 in treatment Period 3; further followed by dose level 7 was planned to receive on Day 1 in treatment Period 4. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7: Participants in Part A Cohort 2 received a single dose of GSK3186899 300 mg on Day 1 in treatment Period 1; followed by a single dose of Placebo on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 800 mg on Day 1 in treatment Period 3; further followed by dose level 7 was planned to receive on Day 1 in treatment Period 4. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended. There was a washout period of 10 days between each treatment period.
- Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7: Participants in Part A Cohort 2 received a single dose of Placebo on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 600 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3186899 800 mg on Day 1 in treatment Period 3; further followed by dose level 7 was planned to receive on Day 1 in treatment Period 4. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended. There was a washout period of 10 days between each treatment period.
- Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed): Participants in Part A Cohort 3 were planned to receive a single dose of GSK3186899 under fasted conditions on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 under fed conditions on Day 1 in treatment Period 2. There was a planned washout period of 10 days between each treatment period.
- Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted): Participants in Part A Cohort 3 were planned to receive a single dose of GSK3186899 under fed conditions on Day 1 in treatment Period 1; followed by a single dose of GSK3186899 under fasted conditions on Day 1 in treatment Period 2. There was a planned washout period of 10 days between each treatment period.
- Part B: Cohort 4- GSK3186899 or Placebo: Participants in Part B Cohort 4 were planned to receive repeat dose of GSK3186899 or placebo on Days 1 to 10.
- Part B: Cohort 5- GSK3186899 or Placebo: Participants in Part B Cohort 5 were planned to receive repeat dose of GSK3186899 or placebo on Days 1 to 10.
- Part B: Cohort 6- GSK3186899 or Placebo: Participants in Part B Cohort 6 were planned to receive repeat dose of GSK3186899 or placebo on Days 1 to 10.
Period: Part A: Cohort 1-Period 1 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod1(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 2 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 | 2 | 2 | 2 (New participant enrolled and dosed) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod2(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 3 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 (New participant enrolled and dosed.) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort1-WashoutPeriod3(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 1-Period 4 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 2 | 2 | 2 | 2 (New participant enrolled and dosed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 1 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized in error | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod1(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 2 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 2 (New participant enrolled and dosed.) | 2 (New participant enrolled and dosed.) | 2 | 2 (New participant enrolled and dosed.) | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod2(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 3 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 2 (New participant enrolled and dosed.) | 2 | 2 (New participant enrolled and dosed.) | 2 | 0 | 0 | 0 | 0 | 0
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort2-WashoutPeriod3(Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 2-Period 4 (Day1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 3- Period 1 (Day 1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA:Cohort3-WashoutPeriod (Upto Day10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort 3- Period 2 (Day 1)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Cohorts 4 to 6 (Days 1 to 10)
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated after completion of Cohort 2, Period 3 of Part A following strategic review after emergence of nonclinical data with non-GlaxoSmithKline asset. Hence, no participants were enrolled in Cohort 2 Period 4 and Cohort 3 of Part A and in all Cohorts of Part B. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1-GSK3186899 30 mg/60 mg/120 mg/Placebo | Part A:Cohort 1-GSK3186899 30 mg/60 mg/Placebo/300 mg | Part A:Cohort 1-GSK3186899 30 mg/Placebo/120 mg/300 mg | Part A:Cohort 1-Placebo/GSK3186899 60 mg/120 mg/300 mg | Part A:Cohort 2-GSK3186899 300 mg/600 mg/800 mg/Placebo | Part A:Cohort 2-GSK3186899 300 mg/600 mg/Placebo/Dose Level 7 | Part A:Cohort 2-GSK3186899 300 mg/Placebo/800 mg/Dose Level 7 | Part A:Cohort 2-Placebo/GSK3186899 600 mg/800 mg/Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo | Total
Number analyzed (Participants) | 3 | 2 | 2 | 4 | 4 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were reported for Safety Population which consisted of all randomized participants who received at least one dose of study treatment.
  Years | 44.7 (6.51) | 34.0 (1.41) | 33.0 (8.49) | 31.3 (8.77) | 34.5 (13.20) | 37.3 (4.04) | 39.7 (8.50) | 41.0 (10.54) |  |  |  |  |  | 36.9 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were reported for Safety Population which consisted of all randomized participants who received at least one dose of study treatment.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 3 | 2 | 2 | 4 | 4 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Baseline characteristics were reported for Safety Population which consisted of all randomized participants who received at least one dose of study treatment.
  Participants
    Asian - Central/South Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian - South East Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    White - White/Caucasian/European Heritage | 3 | 2 | 1 | 3 | 3 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 19
    Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Mixed Race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Non-serious Adverse Events (Non-SAEs) and SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, important medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above. Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to Week 12
Population: Safety Population. Data for Part A: Cohorts 1 and 2- Placebo and Part A: Cohorts 1 and 2- GSK3186899 300 mg arms were presented in a single arm because of similar dosing strategies as pre-defined in the protocol. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohorts 1 and 2- Placebo: Participants in Part A Cohorts 1 and 2 received a single dose of placebo on Day 1 in either treatment Periods 1, 2, 3 and 4.
- Part A: Cohort 1- GSK3186899 30 mg: Participants in Part A Cohort 1 received a single dose of GSK3186899 30 mg on Day 1 in treatment Period 1.
- Part A: Cohort 1- GSK3186899 60 mg: Participants in Part A Cohort 1 received a single dose of GSK3186899 60 mg on Day 1 in treatment Period 2.
- Part A: Cohort 1- GSK3186899 120 mg: Participants in Part A Cohort 1 received a single dose of GSK3186899 120 mg on Day 1 in treatment Period 3.
- Part A: Cohorts 1 and 2- GSK3186899 300 mg: Participants in Part A received a single dose of GSK3186899 300 mg on Day 1 in treatment Period 4 of Cohort 1 and treatment Period 1 of Cohort 2.
- Part A: Cohort 2- GSK3186899 600 mg: Participants in Part A Cohort 2 received a single dose of GSK3186899 600 mg on Day 1 in treatment Period 2.
- Part A: Cohort 2- GSK3186899 800 mg: Participants in Part A Cohort 2 received a single dose of GSK3186899 800 mg on Day 1 in treatment Period 3.
- Part A: Cohort 2- GSK3186899 Dose Level 7: Participants in Part A Cohort 2 were planned to receive dose level 7 on Day 1 in treatment Period 4. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Non-SAEs | 5 | 1 | 2 | 3 | 5 | 2 | 3 |
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

2. Primary Outcome: Part A- Cohort 3: Number of Participants With Non-SAEs and SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, important medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part B: Number of Participants With Non-SAEs and SAEs
Description: as for outcome 2
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: PCI ranges were <0.0 or >0.1*10^9 cells per(/)liter(L)(basophils), <37 or >50 proportion of red blood cells(RBC) in blood(hematocrit),<130 or >170 grams/L(hemoglobin[Hb]), <1.2 or >3.65*10^9cells(c)/L (lymphocytes),<0.2 or >1*10^9c/L(monocytes), <2 or >7.5*10^9c/L(neutrophils), <150 or >400*10^9 c/L(platelets), <3.0 or >10*10^9c/L(white blood cell[WBC]count), <4.4 or >5.8*10^12 c/L(RBC count), <80 or >99 femtoliter(mean corpuscular[MC] volume), <26.0 or >33.5 picogram(MC Hb), <0.0 or >0.4*10^9 c/L(eosinophils). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High) or whose value became within range, were recorded in To within Range or No Change category.Participants were counted twice if participant had values that changed To Low and To High, so the percentages may not add to 100 percentage(%).
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Basophils: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Basophils: To within range or no change | 14 | 6 | 6 | 6 | 12 | 5 | 6 |
  Basophils: To high | 0 | 0 | 0 | 0 | 0 | 1 | 0 |
  Hematocrit: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hematocrit: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Hematocrit: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hemoglobin: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hemoglobin: To within range or no change | 13 | 6 | 6 | 6 | 12 | 6 | 6 |
  Hemoglobin: To high | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Lymphocytes: To low | 2 | 0 | 0 | 0 | 0 | 0 | 0 |
  Lymphocytes: To within range or no change | 12 | 6 | 6 | 6 | 12 | 6 | 6 |
  Lymphocytes: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Monocytes: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Monocytes: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Monocytes: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Neutrophils: To low | 1 | 0 | 0 | 0 | 0 | 1 | 0 |
  Neutrophils: To within range or no change | 12 | 6 | 6 | 6 | 12 | 5 | 6 |
  Neutrophils: To high | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Platelets: To low | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
  Platelets: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 5 |
  Platelets: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  RBC count: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  RBC count: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  RBC count: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  WBC count: To low | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  WBC count: To within range or no change | 12 | 6 | 6 | 6 | 12 | 6 | 6 |
  WBC count: To high | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  MC volume: To low | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
  MC volume: To within range or no change | 13 | 6 | 6 | 6 | 12 | 6 | 5 |
  MC volume: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  MC Hb: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  MC Hb: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  MC Hb: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Eosinophils: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Eosinophils: To within range or no change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Eosinophils: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

5. Primary Outcome: Part A- Cohort 3: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze hematology parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze hematology parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: PCI ranges were <34 or >50 grams/L(albumin),<40 or >129 international units/L[IU/L](alkaline phosphatase),<10 or >50 IU/L(alanine aminotransferase),<0 or >37(aspartate aminotransferase), <0 or >20 micromoles(mcmol)/L (direct bilirubin),<0 or >20 mcmol/L(bilirubin), <2.2 or >2.6 millimoles/L(mmol/L)(calcium),<66 or >112 upper limit of normal mmol/L(creatinine), <3.5 or >5.1 mmol/L (potassium),<0.6 or >1 mmol/L (magnesium),<0.87 or >1.45mmol/L (phosphate),<63 or >83 g/L (protein),<135 or >145 mmol/L (sodium), <0.0 or >5.0 mg/L (C-reactive protein). Participants were counted in worst case category that their value changes to(low, within range [WR] or no change[NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became WR, were recorded in To WR or NC category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Albumin: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Albumin: To within range or NC | 11 | 6 | 6 | 6 | 11 | 6 | 6 |
  Albumin: To high | 3 | 0 | 0 | 0 | 1 | 0 | 0 |
  Alkaline phosphatase: To low | 0 | 0 | 0 | 0 | 2 | 0 | 0 |
  Alkaline phosphatase: To within range or NC | 14 | 6 | 6 | 6 | 10 | 6 | 6 |
  Alkaline phosphatase: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Alanine aminotransferase: To low | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Alanine aminotransferase: To within range or NC | 13 | 6 | 6 | 6 | 12 | 6 | 5 |
  Alanine aminotransferase: To high | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
  Aspartate aminotransferase: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Aspartate aminotransferase: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 5 |
  Aspartate aminotransferase: To high | 0 | 0 | 0 | 0 | 0 | 0 | 1 |
  Direct bilirubin: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Direct bilirubin: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Direct bilirubin: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Bilirubin: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Bilirubin: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Bilirubin: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Calcium: To low | 0 | 0 | 0 | 2 | 0 | 0 | 0 |
  Calcium: To within range or NC | 14 | 6 | 6 | 4 | 12 | 6 | 6 |
  Calcium: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Creatinine: To low | 1 | 0 | 0 | 0 | 0 | 0 | 0 |
  Creatinine: To within range or NC | 13 | 6 | 6 | 6 | 12 | 6 | 6 |
  Creatinine: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Potassium: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Potassium: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Potassium: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Magnesium: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Magnesium: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Magnesium: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Phosphate: To low | 1 | 1 | 1 | 1 | 1 | 0 | 1 |
  Phosphate: To within range or NC | 12 | 4 | 4 | 5 | 11 | 6 | 5 |
  Phosphate: To high | 1 | 1 | 1 | 0 | 0 | 0 | 0 |
  Protein: To low | 1 | 0 | 1 | 0 | 0 | 0 | 0 |
  Protein: To within range or NC | 13 | 6 | 5 | 6 | 12 | 6 | 6 |
  Protein: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Sodium: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Sodium: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Sodium: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  C-reactive protein: To low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  C-reactive protein: To within range or NC | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  C-reactive protein: To high | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

8. Primary Outcome: Part A- Cohort 3: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze chemistry parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Blood samples were planned to be collected to analyze chemistry parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Worst-Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected for analysis of occult blood, ketones and protein by a dipstick method. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine occult blood and protein can be read as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Any increase means any increase to trace, 1+, 2+ or 3+ post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Occult blood | 1 | 0 | 0 | 1 | 0 | 0 | 1 |
  Protein | 2 | 0 | 0 | 0 | 0 | 0 | 1 |
  Ketones | 1 | 1 | 0 | 0 | 0 | 0 | 0 |

11. Primary Outcome: Part A- Cohort 3: Number of Participants With Worst-Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were planned to be collected to analyze urine parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Part B: Number of Participants With Worst-Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were planned to be collected to analyze urine parameters.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT intervals. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Abnormal - not clinically significant | 2 | 1 | 1 | 2 | 4 | 2 | 3 |
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

14. Primary Outcome: Part A- Cohort 3: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings
Description: Twelve lead ECGs were planned to be performed to measure PR interval, QRS duration, QT interval and corrected QT intervals.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Part B: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings
Description: as for outcome 14
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

16. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate, respiratory rate and body temperature and were measured in a semi-supine position after 5 minutes rest. PCI ranges were, SBP (millimeters of mercury [mmHg]): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), pulse rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute): <10(low) or >25(high) and body temperature (degrees Celsius) <35 (low) or >38 (high). Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose vital signs value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  SBP: To Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
  SBP: To within Range or No Change | 14 | 6 | 6 | 5 | 12 | 6 | 6 |
  SBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  DBP: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  DBP: To within Range or No Change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  DBP: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Pulse rate: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Pulse rate: To within Range or No Change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Pulse rate: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Respiratory rate: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Respiratory rate: To within Range or No Change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Respiratory rate: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Body temperature: To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Body temperature: To within Range or No Change | 14 | 6 | 6 | 6 | 12 | 6 | 6 |
  Body temperature: To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

17. Primary Outcome: Part A- Cohort 3: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs were planned to be measured in a semi-supine position after 5 minutes of rest.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Part B: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline
Description: Vital signs were planned to be measured in a semi-supine position after 5 minutes of rest.
Time Frame: Up to Week 9
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

19. Primary Outcome: Part A- Cohorts 1 and 2: Number of Participants With Abnormal Cardiac Telemetry Findings
Description: Continuous cardiac telemetry was performed in a supine position after at least 5 minutes of rest. Abnormal findings were categorized as CS and not NCS. Clinically significant abnormal findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to 24 hours post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 12 | 6 | 6 | 0
Participants
  Abnormal - not clinically significant | 3 | 0 | 3 | 1 | 4 | 2 | 1 |
  Abnormal - clinically significant | 0 | 0 | 1 | 0 | 0 | 0 | 1 |

20. Primary Outcome: Part A- Cohort 3: Number of Participants Abnormal Cardiac Telemetry Findings
Description: Continuous cardiac telemetry was planned to be performed in a supine position after at least 5 minutes of rest.
Time Frame: Up to 24 hours post-dose
Population: Safety Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Part B: Number of Participants Abnormal Cardiac Telemetry Findings
Description: Continuous cardiac telemetry was planned to be performed in a supine position after at least 5 minutes of rest.
Time Frame: Up to 24 hours post-dose
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Part A- Cohorts 1 and 2: Plasma Concentration After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3186899. PK Population consisted of all participants in the Safety Population who received at least 1 non-missing PK assessment.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed. Data for Part A: Cohorts 1 and 2- GSK3186899 300 mg arm was presented in a single arm because of similar dosing strategies as pre-defined in the protocol.Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Nanogram per milliliter
  Pre-dose | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) |
  10 minutes | 36.935 (43.8179) | 10.780 (7.4009) | 68.788 (50.1741) | 183.693 (151.2143) | 528.360 (530.7085) | 766.898 (691.4467) |
  30 minutes | 182.825 (69.0839) | 220.846 (78.8200) | 817.218 (528.0808) | 2112.646 (943.7797) | 5337.077 (1679.9417) | 7563.453 (3748.7402) |
  1 hour | 246.298 (89.0970) | 308.820 (76.3337) | 1217.430 (414.4935) | 2445.121 (846.7178) | 6213.155 (2228.1232) | 8148.812 (3230.8260) |
  1.5 hours | 193.372 (75.7409) | 292.106 (70.6847) | 1165.735 (405.0558) | 2809.873 (731.2502) | 6676.070 (1731.9990) | 7828.908 (1936.6359) |
  2 hours | 169.883 (79.6579) | 266.122 (76.2478) | 1019.690 (317.4601) | 2740.957 (919.9618) | 6388.922 (1338.2507) | 8139.085 (1761.2188) |
  2.5 hours | 143.448 (69.7562) | 296.102 (44.6567) | 981.000 (287.9601) | 2661.372 (869.2819) | 6930.995 (1697.9608) | 7714.882 (2565.6688) |
  3 hours | 124.742 (67.6108) | 297.366 (98.0691) | 841.170 (203.0633) | 2496.468 (751.3136) | 7377.713 (1718.2385) | 8306.098 (2966.1881) |
  4 hours | 71.845 (41.2573) | 211.540 (98.3222) | 586.375 (187.1841) | 2202.511 (908.6908) | 5230.308 (1817.4993) | 6492.033 (2264.4485) |
  5 hours | 48.675 (29.1569) | 149.386 (77.3929) | 407.900 (132.1951) | 1715.797 (818.4628) | 3910.825 (1174.7813) | 5828.517 (1559.1849) |
  6 hours | 33.648 (18.7418) | 109.636 (61.8823) | 318.288 (101.9840) | 1413.953 (714.4323) | 3752.580 (662.1178) | 5010.553 (1424.1685) |
  8 hours | 19.023 (12.4100) | 58.322 (30.3314) | 180.300 (67.3578) | 1008.525 (554.8121) | 3196.830 (1133.3168) | 4352.842 (1510.7803) |
  10 hours | 9.447 (6.7790) | 30.156 (14.0233) | 111.350 (40.8868) | 673.839 (419.1869) | 2571.757 (1287.9872) | 3519.375 (1243.8441) |
  12 hours | 4.975 (3.8146) | 14.662 (9.4905) | 53.978 (33.6205) | 394.246 (259.4013) | 1818.825 (952.8830) | 2676.418 (1366.8170) |
  24 hours | 0.000 (0.0000) | 1.526 (1.0015) | 4.078 (1.2666) | 39.462 (31.0353) | 457.593 (549.4177) | 787.852 (862.1917) |

23. Secondary Outcome: Part A- Cohort 3: Plasma Concentration After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part A- Cohorts 1 and 2: Area Under the Plasma Concentration-time Curve From Time 0 to Last Time of Quantifiable Concentration (AUC[0-t]) After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed. Data for Part A: Cohorts 1 and 2- GSK3186899 300 mg arm was presented in a single arm because of similar dosing strategies as pre-defined in the protocol. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Hours*nanogram per milliliter | 725.40 (41.62) | 1597.85 (32.30) | 5268.31 (31.32) | 18105.45 (47.08) | 58201.67 (29.14) | 77531.24 (34.57) |

25. Secondary Outcome: Part A- Cohort 3: AUC(0-t) After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Part A- Cohorts 1 and 2: Area Under the Plasma Concentration-time Curve From Time 0 to Extrapolated to Infinity (AUC[0-infinity]) After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Hours*nanogram per milliliter | 739.13 (42.31) | 1607.27 (32.10) | 5287.60 (31.20) | 18265.32 (47.50) | 61539.43 (35.59) | 83867.58 (42.98) |

27. Secondary Outcome: Part A- Cohort 3: AUC(0-infinity) After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Part A- Cohorts 1 and 2: Maximum Observed Plasma Drug Concentration (Cmax) After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Nanogram per milliliter | 239.206 (34.38) | 356.232 (19.32) | 1214.000 (29.72) | 3011.334 (37.57) | 8219.997 (15.50) | 9445.301 (28.78) |

29. Secondary Outcome: Part A- Cohort 3: Cmax After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Part A- Cohorts 1 and 2: Time to Maximum Observed Plasma Drug Concentration (Tmax) After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 24
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Hour | 1.00 [0.5 to 1.5] | 3.00 [1.0 to 3.0] | 1.00 [1.0 to 1.5] | 2.00 [1.0 to 4.0] | 2.75 [1.0 to 3.0] | 2.50 [1.0 to 4.0] |

31. Secondary Outcome: Part A- Cohort 3: Tmax After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Part A- Cohorts 1 and 2: Trough Plasma Concentration (Ctau) After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected for this endpoint as it was incorrectly stated as one of the Secondary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to Ctau for single ascending dose part was an error. Data for Part A: Cohorts 1 and 2- GSK3186899 300 mg arm was planned to be presented in a single arm because of similar dosing strategies as pre-defined in the protocol.
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Part A- Cohort 3: Ctau After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Part A- Cohorts 1 and 2: Apparent Terminal Half-life (T1/2) After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 24
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Hour | 1.982 [1.44 to 2.44] | 2.955 [1.66 to 3.50] | 2.758 [2.58 to 3.93] | 3.302 [2.65 to 3.98] | 4.655 [3.22 to 8.93] | 5.135 [4.32 to 10.78] |

35. Secondary Outcome: Part A- Cohort 3: T1/2 After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part A- Cohorts 1 and 2: Predicted Accumulation Ratio After Single Dose Administration of GSK3186899
Description: Blood samples were collected at indicated time points for PK analysis of GSK3186899. Predicted accumulation ratio is calculated as 1/(1-e^[k*tau]) where k is elimination rate constant following the single dose and tau is the dosing interval for the intended repeat dosing.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7
Number analyzed (Participants) | 6 | 5 | 4 | 10 | 6 | 6 | 0
Ratio | 1.0183 (0.01324) | 1.0631 (0.03952) | 1.0704 (0.04505) | 1.0889 (0.03246) | 1.2603 (0.19948) | 1.3429 (0.26138) |

37. Secondary Outcome: Part A- Cohort 3: Predicted Accumulation Ratio After Single Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Part B: Plasma Concentration After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: Days 1 and 10: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose; Days 2 to 9: Pre-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

39. Secondary Outcome: Part B: AUC(0-t) After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Part B: AUC(0-infinity) After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Part B: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval (AUC[0-tau]) After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

42. Secondary Outcome: Part B: Cmax After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Part B: Tmax After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

44. Secondary Outcome: Part B: T1/2 After Repeat Dose Administration of GSK3186899
Description: Blood samples were planned to be collected at indicated time points for PK analysis of GSK3186899.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

45. Secondary Outcome: Part A- Cohorts 1 and 2: Dose-proportionality of GSK3186899 Administered as Single Dose Based on AUC(0-infinity)
Description: Blood samples were collected at indicated time points for PK analysis. Dose proportionality was assessed using Power model with fixed effects of logarithm of treatment and participant as random effect. Slope and 90% confidence interval for the slope are presented.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Only those participants with data available at the specified time points were analyzed. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as the stopping criteria was reached with the 800mg dose and no further dose escalation was recommended.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part A: Cohorts 1 and 2- GSK3186899 30 to 800 mg: Participants in Part A received a single dose of GSK3186899 30, 60, 120, 300, 600 and 800 mg in any of the treatment Periods of Cohorts 1 or 2 according to randomization schedule.
Arm/Group | Part A: Cohorts 1 and 2- GSK3186899 30 to 800 mg
Number analyzed (Participants) | 22
Slope of log dose | 1.47 [1.34 to 1.61]

46. Secondary Outcome: Part A- Cohort 3: Dose-proportionality of GSK3186899 Administered as Single Dose Based on AUC(0-infinity)
Description: Blood samples were planned to be collected at indicated time points for PK analysis.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Part A- Cohorts 1 and 2: Dose-proportionality of GSK3186899 Administered as Single Dose Based on Cmax
Description: as for outcome 45
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: as for outcome 45
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Part A: Cohorts 1 and 2- GSK3186899 30 to 800 mg
Number analyzed (Participants) | 22
Slope of log dose | 1.19 [1.09 to 1.30]

48. Secondary Outcome: Part A- Cohort 3: Dose-proportionality of GSK3186899 Administered as Single Dose Based on Cmax
Description: Blood samples were planned to be collected at indicated time points for PK analysis.
Time Frame: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose in each treatment period
Population: PK Population. Data was not collected as no participants were enrolled in Part A Cohort 3.
Arm/Group | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted)
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Part B: Dose-proportionality of GSK3186899 Administered as Repeat Dose Based on AUC(0-tau)
Description: Blood samples were planned to be collected at indicated time points for PK analysis.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

50. Secondary Outcome: Part B: Dose-proportionality of GSK3186899 Administered as Repeat Dose Based on Cmax
Description: Blood samples were planned to be collected at indicated time points for PK analysis.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

51. Secondary Outcome: Part B: Dose-proportionality of GSK3186899 Administered as Repeat Dose Based on Ctau
Description: Blood samples were planned to be collected at indicated time points for PK analysis.
Time Frame: as for outcome 38
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

52. Secondary Outcome: Part B: Relative Accumulation Ratio of GSK3186899 After Repeat Dose Administration by AUC(0-tau)
Description: Blood samples were planned to be collected at indicated time points for PK analysis. Accumulation ratio was planned to be calculated as ratio of AUC(0-tau) at Day 10 to AUC(0-tau) at Day 1.
Time Frame: Days 1 and 10: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

53. Secondary Outcome: Part B: Relative Accumulation Ratio of GSK3186899 After Repeat Dose Administration by Cmax
Description: Blood samples were planned to be collected at indicated time points for PK analysis. Accumulation ratio was planned to be calculated as ratio of Cmax at Day 10 to Cmax at Day 1.
Time Frame: Days 1 and 10: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

54. Secondary Outcome: Part B: Relative Accumulation Ratio of GSK3186899 After Repeat Dose Administration by Ctau
Description: Blood samples were planned to be collected at indicated time points for PK analysis. Accumulation ratio was planned to be calculated as ratio of Ctau at Day 10 to Ctau at Day 1.
Time Frame: Days 1 and 10: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

55. Secondary Outcome: Part B: Time Invariance Ratio of GSK3186899 After Repeat Dose Administration Using AUC
Description: Blood samples were planned to be collected at indicated time points for PK analysis. Time-invariance ratio was planned to be calculated as AUC(0-12) on Day 10 to AUC(0-infinity) on Day 1.
Time Frame: Days 1 and 10: Pre-dose, 10, 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, and 12 hours post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-SAE and SAE were collected up to Week 12 in Part A. Data for Part A: Cohorts 1 and 2- Placebo and Part A: Cohorts 1 and 2- GSK3186899 300 mg arms were presented in a single arm because of similar dosing strategies as pre-defined in the protocol. Dose level 7 was not conducted as dose escalation was stopped at dose level 6 (800 mg), as stopping criteria was reached with 800 mg dose and no further dose escalation was recommended.
Description: All-cause mortality,non-SAE,SAE were collected using Safety Population in Cohorts1and2 of PartA.1 participant from Enrolled Population(N=25) did not receive study treatment,hence was not included in Safety Population(N=24).Data was not collected in Cohort2-Period4,Cohort3 of PartA and PartB as study was terminated and no participant was enrolled in these cohorts/parts.
Arm/Group | Part A: Cohorts 1 and 2- Placebo | Part A: Cohort 1- GSK3186899 30 mg | Part A: Cohort 1- GSK3186899 60 mg | Part A: Cohort 1- GSK3186899 120 mg | Part A: Cohorts 1 and 2- GSK3186899 300 mg | Part A: Cohort 2- GSK3186899 600 mg | Part A: Cohort 2- GSK3186899 800 mg | Part A: Cohort 2- GSK3186899 Dose Level 7 | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) | Part B: Cohort 4- GSK3186899 or Placebo | Part B: Cohort 5- GSK3186899 or Placebo | Part B: Cohort 6- GSK3186899 or Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/14 | 1/6 | 2/6 | 3/6 | 5/12 | 2/6 | 3/6 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohorts 1 and 2- Placebo (N=14) | Part A: Cohort 1- GSK3186899 30 mg (N=6) | Part A: Cohort 1- GSK3186899 60 mg (N=6) | Part A: Cohort 1- GSK3186899 120 mg (N=6) | Part A: Cohorts 1 and 2- GSK3186899 300 mg (N=12) | Part A: Cohort 2- GSK3186899 600 mg (N=6) | Part A: Cohort 2- GSK3186899 800 mg (N=6) | Part A: Cohort 2- GSK3186899 Dose Level 7 (N=0) | Part A: Cohort 3- GSK3186899 (Fasted) + GSK3186899 (Fed) (N=0) | Part A: Cohort 3- GSK3186899 (Fed) + GSK3186899 (Fasted) (N=0) | Part B: Cohort 4- GSK3186899 or Placebo (N=0) | Part B: Cohort 5- GSK3186899 or Placebo (N=0) | Part B: Cohort 6- GSK3186899 or Placebo (N=0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03874234/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03874234/SAP_001.pdf